CLINICAL TRIAL: NCT02484560
Title: Efficacy of Allogenic Mesenchymal Stem Cell Therapy in Ambulatory and Non-ambulatory Children With Duchenne Muscular Dystrophy - Phase 1-2
Brief Title: Efficacy of Stem Cell Therapy in Ambulatory and Non-ambulatory Children With Duchenne Muscular Dystrophy - Phase 1-2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Gaziantep (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, Alper Dai, MD, Lead Investigator, University of Gaziantep
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56733164/203
Record Dates: First submitted 2015-06-16; First posted 2015-06-29 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Neuromuscular Diseases; Muscular Dystrophy; Genetic Diseases, X-linked; Musculoskeletal Diseases; Nervous System Diseases
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Neuromuscular Diseases; Muscular Dystrophies; Genetic Diseases, X-Linked; Musculoskeletal Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambulatory Patients (Experimental): Ambulatory patients receiving stem cell therapy
  Interventions: Drug: Biological: Umbilical Cord Based Allogenic Mesenchymal Stem Cell
- Non-Ambulatory Patients (Experimental): non-ambulatory patients receiving stem cell therapy
  Interventions: Drug: Biological: Umbilical Cord Based Allogenic Mesenchymal Stem Cell

INTERVENTIONS:
Drug: Biological: Umbilical Cord Based Allogenic Mesenchymal Stem Cell

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is a X-linked genetic disorder primarily affecting males, resulting in an absence of dystrophin which ultimately leads to progressive muscle degeneration. Patients with DMD progressively lose functional abilities of movement, breath, and eventually the ability to circulate blood. Currently, there is no cure for DMD, although several strategies are being tested for treatment, none have yet proven to be sufficient. Children with DMD are generally divided into two groups based on severity or progression of the disease, non-ambulatory and ambulatory. Ambulatory patients are capable of walking independently while non-ambulatory patients cannot walk independently.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is a X-linked genetic disorder primarily affecting males, resulting in an absence of dystrophin which ultimately leads to progressive muscle degeneration. Patients with DMD progressively lose functional abilities of movement, breath, and eventually the ability to circulate blood. Currently, there is no cure for DMD, although several strategies are being tested for treatment, none have yet proven to be sufficient. Children with DMD are generally divided into two groups based on severity or progression of the disease, non-ambulatory and ambulatory. Ambulatory patients are capable of walking independently while non-ambulatory patients cannot walk independently.

The purpose of this study is to investigate the effects of Allogenic Mesenchymal Stem Cell Therapy in Ambulatory and Non-ambulatory Children with Duchenne Muscular Dystrophy and determine its suitability as a form of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory and Non-ambulatory patients diagnosed with DMD that is proven both clinically and genetically and are between 5-20 years old who need partial respiratory support daily. Patients with less than or equal to stage 1 NIH, cardiac, liver, and renal function. Patients must also not present any indication of cancer, allergic disease, nor bleeding diathesis.

Exclusion Criteria:

* Patients who require full respiratory support. Patients have stage II NIH or greater, cardiac, liver, and renal function. Patients present with signs of symptoms of cancer, allergic disease, or bleeding diathesis.

Ages: 8 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Degree of improvement in patients with Duchenne Muscular Dystrophy after stem cell therapy treatment administered using Northstar Ambulatory Assessment, Magnetic Resonance Imaging & Spectroscopy, muscle strength assessment equipment, and a questionnaire. | 12 Months
  Tests Used in Assement:
  Northstar ambulatory assessment CHAQ (Child Health Assessment Questionnaire) MRI/MRS Muscle Strength Assessment - Myogrip, Myopinch, and Moviplate

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University Hospital, Gaziantep, Turkey (Türkiye)